CLINICAL TRIAL: NCT05681325
Title: Evaluation of Antioxidant and Anti-inflammatory Effect of Matcha Tea Intake on Periodontal Health
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hayder Raad Abdulbaqi (Other)
Responsible Party: Sponsor-Investigator, Hayder Raad Abdulbaqi, professor, University of Baghdad
Organization: University of Baghdad (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: matcha on periodontal health
Record Dates: First submitted 2022-12-11; First posted 2023-01-12 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Gingival Disease
MeSH Terms: conditions — Gingival Diseases | interventions — Tea

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- green tea group (Active Comparator): Mahmood Green Tea Sri Lanka. It will be given 2 cups / day for 30 days.
  Interventions: Dietary Supplement: green tea
- matcha tea group (Experimental): Jade Leaf Organic Japanese Matcha, USA. It will be given 2 cups / day for 30 days.
  Interventions: Dietary Supplement: matcha tea

INTERVENTIONS:
Dietary Supplement: green tea — It will be given 2 cups / day for 30 days. To prepare each cup, a tea pack will be immersed into a cup of hot water.
  Arms: green tea group
Dietary Supplement: matcha tea — It will be given 2 cups / day for 30 days. To prepare each cup, a tea pack will be immersed into a cup of hot water.
  Arms: matcha tea group

SUMMARY:
Aim of the study:

This study aims to evaluate the antioxidant and beneficial effects of matcha tea daily intake on periodontal health.

Objectives:

* To evaluate the salivary level of antioxidants (catalase, total antioxidant capacity) after matcha tea intake compared to green tea over a period of one month.
* To evaluate the clinical periodontal parameters including bleeding on probing (BOP), probing pocket depth (PPD) and plaque index (PI) after matcha tea intake compared to green tea over a period of one month.
* To evaluate the salivary levels of IL-1B after matcha tea intake compared to green tea over a period of one month.

ELIGIBILITY:
Inclusion Criteria:

* • having at least 20 teeth,

  * underwent no medical treatment during the last 3 months before examination and sampling,
  * non-smoker,
  * no history of systemic disease,
  * gingivitis patient (having >10% bleeding sites with no PPD >3 mm).

Exclusion Criteria:

* • wore orthodontic appliances,

  * pregnant or currently in the breast-feeding period,
  * periodontitis patient,
  * smoker,
  * has a history of systemic disease.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-01-25 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-07-12 (Estimated)

PRIMARY OUTCOMES:
change in salivary level of antioxidant marker | 30 Days (baseline to one moth of tea intake)
  change in level of catalase enzyme in ku/L
change in salivary level of ant-inflammatory marker | 30 Days (baseline to one moth of tea intake)
  change in level of interleukin- one beta (IL-1B) in pg/L

SECONDARY OUTCOMES:
change in percentage of bleeding on probing (BOP) | 30 Days (baseline to one moth of tea intake)
  change in BOP percentage. less percentage means less inflammation in gingival tissue
change in plaque index (PI) scores | 30 Days (baseline to one moth of tea intake)
  change in PI scores. less scores mean less dental plaque accumulated onto teeth surfaces

CONTACTS AND LOCATIONS:
Overall Officials: HIND KAREEM, BDS, Study Director — University of Baghdad
Locations (1):
- Universality of Baghdad, College of dentistry, Baghdad, Iraq

REFERENCES:
- [Background] Zhang Y, Kang N, Xue F, Qiao J, Duan J, Chen F, Cai Y. Evaluation of salivary biomarkers for the diagnosis of periodontitis. BMC Oral Health. 2021 May 17;21(1):266. doi: 10.1186/s12903-021-01600-5. PMID 34001101
- [Background] Kolackova T, Kolofikova K, Sytarova I, Snopek L, Sumczynski D, Orsavova J. Matcha Tea: Analysis of Nutritional Composition, Phenolics and Antioxidant Activity. Plant Foods Hum Nutr. 2020 Mar;75(1):48-53. doi: 10.1007/s11130-019-00777-z. PMID 31832980